CLINICAL TRIAL: NCT01262313
Title: Healthy Creations: Community Based Lifestyle Intervention Validation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GFHNRC019
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Sham Comparator): The Control group will have an hour-long meeting of instruction by a registered dietitian on using the provided "A Healthier You: Everyday Healthy Eating and Physical Activity for Life" book, based on the Dietary Guidelines for Americans 2005.
  Interventions: Behavioral: Lifestyle Counseling
- lifestyle counseling intervention (Experimental): This group will participate in the weekly "Healthy Creations" classes for 8 weeks presented by a Registered Dietitian and a certified fitness trainer. This is a community based lifestyle intervention program.
  Interventions: Behavioral: Lifestyle Counseling

INTERVENTIONS:
Behavioral: Lifestyle Counseling — Participants in the intervention group will attend an 8-week group intervention discussing "Healthy Creations" lifestyle changes.

SUMMARY:
There remain important barriers to the translation of the programs like the Diabetes Prevention Program to public health. There is a lack of established lifestyle intervention programs as they are resource and time intensive, exceeding both the resources and the training of most primary care providers. A solution may be the implementation of lifestyle intervention programs in the community setting that are unrelated to primary medical care. A community based program at a public facility may extend the reach of lifestyle intervention to those unable to obtain these services from an established medical facility. Community lifestyle intervention to modify dietary, physical activity, and behavioral factors may be a promising strategy for weight management and the reduction of risk for metabolic disease. In this validation study we will assess pre and post intervention to identify whether measurable changes can be detected in body weight, body composition, markers of metabolic disease and quality of life after participation in the "Healthy Creations", a community based lifestyle intervention program presented by Center Court Fitness Center of the Grand Forks Park District and Altru Health System.

ELIGIBILITY:
Inclusion Criteria:

* overweight or Class I and II obese
* live in Grand Forks, ND area

Exclusion Criteria:

* history of eating disorder
* pregnancy
* inability to understand English or give consent
* uncontrolled medical condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-12; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Percentage weight change from baseline | 20 weeks
  Participants in the intervention group will attend an 8-week group intervention of "Healthy Creations. Participants in the control group will participate in one class on diet and physical activity presented by a dietitian.

SECONDARY OUTCOMES:
functional fitness | 20 weeks
  Functional fitness will be measured by a 6-minute walk test (cardio-respiratory fitness). Leg strength, core strength, upper body strength, flexibility, and balance will be measured.
insulin sensitivity | 20 weeks
  Changes in insulin sensitivity will be examined using a fasting blood draw.
Plasma Lipids | 20 weeks
  Plasma lipids will be examined using fasting blood draws

CONTACTS AND LOCATIONS:
Overall Officials: Susan K Raatz, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

REFERENCES:
- [Background] Look AHEAD Research Group; Wing RR. Long-term effects of a lifestyle intervention on weight and cardiovascular risk factors in individuals with type 2 diabetes mellitus: four-year results of the Look AHEAD trial. Arch Intern Med. 2010 Sep 27;170(17):1566-75. doi: 10.1001/archinternmed.2010.334. PMID 20876408
- [Background] Raatz SK, Wimmer JK, Kwong CA, Sibley SD. Intensive diet instruction by registered dietitians improves weight-loss success. J Am Diet Assoc. 2008 Jan;108(1):110-3. doi: 10.1016/j.jada.2007.10.010. PMID 18155995
- [Background] Williamson DA, Rejeski J, Lang W, Van Dorsten B, Fabricatore AN, Toledo K; Look AHEAD Research Group. Impact of a weight management program on health-related quality of life in overweight adults with type 2 diabetes. Arch Intern Med. 2009 Jan 26;169(2):163-71. doi: 10.1001/archinternmed.2008.544. PMID 19171813
- [Background] Jakicic JM, Jaramillo SA, Balasubramanyam A, Bancroft B, Curtis JM, Mathews A, Pereira M, Regensteiner JG, Ribisl PM; Look AHEAD Study Group. Effect of a lifestyle intervention on change in cardiorespiratory fitness in adults with type 2 diabetes: results from the Look AHEAD Study. Int J Obes (Lond). 2009 Mar;33(3):305-16. doi: 10.1038/ijo.2008.280. Epub 2009 Jan 20. PMID 19153582